CLINICAL TRIAL: NCT04661670
Title: Relief of Signs and Symptoms in Patients With Tempro-mandibular Disorders Using Occlusal Stabilization Splints Equilibrated by T-scan Versus Articulating Paper: A Randomized Clinical Trial
Brief Title: Occlusal Stabilization Splints Equilibrated by Different Techniques and Their Effect on TMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Eman Saad el Din, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO341
Record Dates: First submitted 2020-12-01; First posted 2020-12-10 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Temporomandibular Joint Disorders
Keywords: equilbration; T scan; Occlusal splints
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor and statistician will be blinded. It is not possible to blind neither the participant nor the care provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- occlusal stabilization splints equilibrated by articulating paper (Active Comparator): In this group the final occlusal correction will be performed with the patient in supine position using 20 um thick articulating paper and articulating foil 8 um thick. The patient will be asked to tap 3 times on the articulating paper and occlusal correction will be done using carbide laboratory bur and rubber cone till uniform contact on all teeth is achieved in centric relation which is illustrated on the splint by a series of uniformly appearing articulating paper dots. Then the patient will be asked to make protrusive and right and left excursions to ensure smooth anterior guidance and posterior disocclusion.
  Interventions: Device: occlusal stabilization splints
- occlusal stabilization splints equilibrated by T-scan (Active Comparator): In this group the same adjustment sequence will be done using T Scan III (software version 8.0) computerized occlusal analysis, a new patient file will be opened, the patient's biological data will be entered, and the T Scan dental arch size is customized to fit the patients arch anatomy. The patient will be asked to clench to record occlusal force and areas that needs adjustment will be grinded using the paper marks as the guideline and carbide laboratory bur till bilateral force balance achieved and the center of force (COF) icon sits close to the midline.
  Mandibular excursions are then adjusted in a similar fashion. Contacts rather than anterior and canine guidance will be eliminated till achieving anterior guidance and posterior disocclusion in time less than 0.5 seconds.
  Interventions: Device: occlusal stabilization splints

INTERVENTIONS:
Device: occlusal stabilization splints — an intraoral appliance that has flat surface to allow bilateral posterior contacts in coincidence with physiologic condylar seating and to produce smooth anterior guidance in excursions
  Other Names: Michigan splint, turner splint

SUMMARY:
The objective of the study is to evaluate if occlusal stabilization splints equilibrated by articulating paper will have equivalent effect in comparison to occlusal stabilization splints equilibrated by T-scan regarding the relief of the TMD signs and symptoms

DETAILED DESCRIPTION:
Eligible patient will be selected from Outpatient Clinic in Prosthodontics Department clinic. Patients will be informed of the nature of the research work and informed consent will be obtained from each of them.All patients will be assessed for TMJ health following DC/TMD Axis I and II to confirm the diagnosis . Base line pain scale and range of pain free jaw movements (mm) will be recorded before starting the treatment. Patients will be randomly divided into 2 equal groups; occlusal stabilization splints equilibrated by articulating paper and occlusal stabilization splints equilibrated by T-scan

Patients of both groups will be subjected to:

Primary impressions will be taken using rubber base impression material (Zhermac zetaplus impression material) ,the impressions will be poured twice to construct 2 study casts to be used for final occlusal adjustment of the splint. Maxillary Face-bow record will be done to mount both maxillary casts on a semi adjustable articulator (A7-Plus Bio Art semi-adjustable articulator) using different mounting rings.

Bite registration using bite registration material (Futar D Bite Registration Material - Ultra Rigid from Kettenbach LP ) will be done in centric relation after deprogramming the muscles using acrylic jig or leaf gauges, followed by loading test for condyle position verification 7to mount the mandibular cast. A protrusive record will be made at 6 mm mandibular protrusion to set the horizontal condylar guidance, while lateral condylar guidance will be adjusted at fixed value of 15 degrees.

The centric relation will be verified by comparing the first point of contact intraorally and the first point of contact on the articulator will be verified. The maxillary cast will be surveyed to detect teeth height of contour. The borders of the occlusal splint will be drawn on the maxillary cast to be occlusal to the height of contour buccally and to extend 1-2 mm beyond the gingival margin on the palatal surface. As the jaw relation and mounting will be done by leaf gauges and at elevated vertical dimension, the incisal pin will be kept on zero. The appliance will be waxed up by filling the inter-arch space with pink wax placed will taper it to a feather edge to the previously drawn borders. A complete arch coverage design will be done and will be shaped to be flat. The wax will be checked with 20 um thick articulating paper (AccuFilm, parkell, USA)and should produce bilateral posterior contacts in coincidence with physiologic condylar seating and a smooth anterior guidance in excursions allowing posterior disocclusion2

A mould for the shaped wax will be done using Polyvinyl silicone elastomer putty material (elite P&P, Italy) in a plastic container. A white self-cured acrylic resin (Acrostone cold cure material) will be mixed and filled inside the mould and will be closed tightly till all excess comes out. After material setting the acrylic occlusal splint will be finished and seated on the duplicated cast and final fit and occlusal correction using 20 um thick articulating paper (AccuFilm, parkell, USA) will be done.

In the next clinical visit the splint will be inserted inside patient's mouth and will be checked for stability and comfort before any occlusal adjustment which will be performed by articulating paper or T-Scan according to the assigned groups.

Study group:

In this group the final occlusal correction will be performed with the patient in supine position using 20 um thick articulating paper (AccuFilm, parkell, USA) and articulating foil (DENU shim stock, HDI) 8 um thick. The patient will be asked to tap 3 times on the articulating paper and occlusal correction will be done using carbide laboratory bur and rubber cone till uniform contact on all teeth is achieved in centric relation which is illustrated on the splint by a series of uniformly appearing articulating paper dots. Then the patient will be asked to make protrusive and right and left excursions to ensure smooth anterior guidance and posterior disocclusion.

Control group:

In this group the same adjustment sequence will be done using T Scan III (software version 8.0) computerized occlusal analysis, a new patient file will be opened, the patient's biological data will be entered, and the T Scan dental arch size is customized to fit the patients arch anatomy. A centric occlusion scan label with Turbo mode (0.003 second incremental scanning) scan speed will be selected. The sensor will be placed intraorally so that the midline 'V' of the support contacts the midline of the occlusal splint. The patient is then asked to gently close on their posterior teeth, then clench firmly against the occlusal splint for one to three seconds. The sensitivity level will be adjusted to fit the patient's occlusal strength. When the sensitivity is properly set, the patient will be asked to clench

to record occlusal force and areas that needs adjustment will be grinded using the paper marks as the guideline and carbide laboratory bur till bilateral force balance achieved and the center of force (COF) icon sits close to the midline.

Mandibular excursions are then adjusted in a similar fashion. The appropriate excursion scan label will be chosen, after which the patient is asked to clench on their posterior teeth for one to three seconds, and then move in a lateral or protrusive excursion to the full extent of the border movement. Contacts rather than anterior and canine guidance will be eliminated till achieving anterior guidance and posterior disocclusion in time less than 0.5 seconds.

For both groups:

After occlusal adjustment in centric relation, the occlusion will be evaluated in upright position and will ensure that patient bites comfortably and that all teeth contact evenly, with no anterior teeth contacting harder than the posterior teeth. No polishing will be done after adjustment for maintenance of the refined occlusal contacts. The patients will be instructed to wear the occlusal splint at nighttime, to alleviate daytime harmful habits, the patients will be instructed to seal the lips and separate the teeth, keeping the muscles relaxed. The patients will be recalled every after 1 week and every 2 weeks for further needed occlusal adjustment till there is no change at all between visits

After 1 month and 3 months, the patients will be recalled to evaluate the improvements in TMD pain symptoms using questionnaires, in addition to the improvement in range of pain free jaw movements using mm ruler.

ELIGIBILITY:
Inclusion Criteria:

1. Adult cooperative patients who have bruxism and TMD of myogenous origin (Age: 18-60)
2. Fully dentate or partial edentulous patients with no more than one missing tooth per quadrant, excluding third molars
3. presence of signs and symptoms of TMD ( diffuse pain in head and neck, headache pain exaggeration by jaw movements, restricted jaw movements)
4. severe Disc displacement with or without reduction who can be treated by stabilization appliance (Reciprocal click, or without click)

   Exclusion Criteria:
5. Use of removable dentures
6. More than one absent tooth per quadrant
7. Patients with anterior open bite
8. Severe systemic conditions or somatic symptoms, depression and anxiety
9. Trauma of recent date towards face, head or neck
10. Dentoalveolar pathology or ongoing treatment related to TMD.
11. patients scheduled for dental procedures that could alter the occlusion during therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Relief of TMD Signs and symptoms | 3 months
  Graded pain scale questionnaire (VAS scale)
Increased range of painless jaw movements | 3 months
  Jaw functional questionnaire (VAS scale)

SECONDARY OUTCOMES:
measurement of range of jaw movements (maximum un assisted opening , protruion, right and left excrusion) | 3 months
  ruler measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf emil, PhD, Study Director — Cairo University; Mohamed Khashab, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Patient1s contact and pre and post data about pain level and jaw movements
Supporting Information: SAP
Time Frame: After 2 years
Access Criteria: a request will be send to me by mail to send the IPD Data

REFERENCES:
- [Background] Kerstein RB, Radke J. Clinician accuracy when subjectively interpreting articulating paper markings. Cranio. 2014 Jan;32(1):13-23. doi: 10.1179/0886963413Z.0000000001. PMID 24660642
- [Background] Garrido Garcia VC, Garcia Cartagena A, Gonzalez Sequeros O. Evaluation of occlusal contacts in maximum intercuspation using the T-Scan system. J Oral Rehabil. 1997 Dec;24(12):899-903. doi: 10.1046/j.1365-2842.1997.00586.x. PMID 9467991